CLINICAL TRIAL: NCT06530160
Title: Comparison Between Leukodepleted and Non-Leukodepleted Packed Red Blood Cells in Interleukin-8 Level as an Inflammatory Cytokine
Brief Title: Interleukin-8 Level in Packed Red Blood Cells
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Wesam Ashraf Soliman Ahmed, Resident doctor, Assiut University
Other Study IDs: Interleukin-8 in packed Rbcs
Record Dates: First submitted 2024-07-27; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Packed Red Blood Cells
Keywords: Interleukin-8
MeSH Terms: interventions — Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ELISA — Enzyme-linked immunosorbent assay

SUMMARY:
1. To compare level of interleukin-8 between leukodepleted and non-leukodepleted packed red blood cells.
2. To show the effect of filtration of packed red blood cells on the level of inflammatory interleukin-8.

DETAILED DESCRIPTION:
The term cytokine was proposed by Stanley Cohen in 1974 and refers to peptides, proteins, and glycoproteins which play a role in controlling the survival/death of cells, their growth and differentiation as well as the effector functions in tissues and immune cells.

The cytokines are small cell-signaling protein molecules with several functions,e.g.: Intracrine, Autocrine and Intercrine actions (1).

They are synthesized by different immune cells, mainly by T cells, neutrophils and macrophages, which are responsible to promote and regulate immune response (i.e. activity, differentiation, proliferation and production of cells and other cytokines) (2).

Cytokines are described as being pro-inflammatory or antiinflammatory, both of which accumulate in blood products during storage mainly as a result of damaged leucocytes. The accumulation of pro-inflammatory cytokines, is regarded as one of the major causative factors For Transfusion-Associated Adverse Reactions (TAARs), particularly Febrile Non-Haemolytic Transfusion Reactions (FNHTRs) and Transfusion-Related Immunomodulation (TRIM). In addition, the transfusion of blood products containing cytokines has been associated with transfusion-induced systemic inflammation in patients with pre-activated endothelial cells (3).

Interleukin-8 (also known as neutrophil-activating peptide 1) is recognized as a potent effector of neutrophil functions. Several different cell types that contact blood, namely T lymphocytes, monocytes, and endothelial cells, secrete this polypeptide following stimulation by cytokines, or lipopolysaccharide (4).

Interleukin-8 (IL-8), a cytokine with chemotactic and activating properties for neutrophils, has recently been isolated, cloned, and expressed.5 IL-8 is produced by monocytes in response to lipopolysaccharide (LPS), tumor necrosis factor-α (TNF-α), and IL-1;6 and has been implicated in the pathogenesis of acute lung injury. Therefore, we hypothesized that IL-8 may be a mediator of the pathologic events in hemolytic transfusion reaction (HTR), and designed an in vitro model of red blood cell (RBC) incompatibility to investigate the possible role of IL-8 in this setting (5).

Leukoreduction (LR) is a potential means of preventing cytokine production (6).

Thus reducing the white blood cell (WBC) content (leukodepletion) in cellular blood components to a significant level has a direct impact on reducing the incidence of many adverse effects of transfusion-associated with leukocytes and cytokines present in higher levels in non leukodepleted blood component (7).

ELIGIBILITY:
Inclusion Criteria:

* In total, 82 donors fulfilling all general criteria for blood donation, different blood groups and socioeconomic backgrounds, males and females belonging to this geographical area.

Exclusion Criteria:

* Donors not fulfilling all general criteria for blood donation according to World Health Organization:
* Age between 18 and 65
* Weight at least 50 kg
* Haemoglobin not less than 13 g/dl in males and 12 g/dl in females
* must be in good health at the time of donation
* Cannot donate if have a cold, flu, sore throat, cold sore, stomach bug or any other infection.
* Have ever had a positive test for HIV (AIDS virus)
* It is not advisable to donate blood while Breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy donors
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Compare level of interleukin-8 between leukodepleted and non-leukodepleted packed red blood cells | Baseline
  Show the effect of filteration of packed red blood cells on the level of inflammatory interleukin-8

REFERENCES:
- [Background] Anaya JM, Shoenfeld Y, Rojas-Villarraga A, Levy RA, Cervera R, editors. Autoimmunity: From Bench to Bedside [Internet]. Bogota (Colombia): El Rosario University Press; 2013 Jul 18. Available from http://www.ncbi.nlm.nih.gov/books/NBK459447/ PMID 29087650
- [Background] Turner MD, Nedjai B, Hurst T, Pennington DJ. Cytokines and chemokines: At the crossroads of cell signalling and inflammatory disease. Biochim Biophys Acta. 2014 Nov;1843(11):2563-2582. doi: 10.1016/j.bbamcr.2014.05.014. Epub 2014 Jun 2. PMID 24892271
- [Background] Darbonne WC, Rice GC, Mohler MA, Apple T, Hebert CA, Valente AJ, Baker JB. Red blood cells are a sink for interleukin 8, a leukocyte chemotaxin. J Clin Invest. 1991 Oct;88(4):1362-9. doi: 10.1172/JCI115442. PMID 1918386
- [Background] Davenport RD, Strieter RM, Standiford TJ, Kunkel SL. Interleukin-8 production in red blood cell incompatibility. Blood. 1990 Dec 15;76(12):2439-42. PMID 1702325
- [Background] Shukla R, Patel T, Gupte S. Release of cytokines in stored whole blood and red cell concentrate: Effect of leukoreduction. Asian J Transfus Sci. 2015 Jul-Dec;9(2):145-9. doi: 10.4103/0973-6247.162708. PMID 26420933